CLINICAL TRIAL: NCT00988286
Title: Mechanism of Action of Biofeedback Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5R01DK057100 (NIH)
Record Dates: First submitted 2009-09-22; First posted 2009-10-02 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: Constipation; Hyposensitivity; Hypersensitivity
MeSH Terms: conditions — Constipation; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CEP (Experimental)
  Interventions: Procedure: CEP, MEP, TMS

INTERVENTIONS:
Procedure: CEP, MEP, TMS — Patients and healthy volunteers will undergo cortical evoked potentials (CEP), motor evoked potentials (MEP) and transcranial evoked potentials (TMS).

SUMMARY:
Biofeedback therapy improves bowel symptoms and anorectal function in patients with dyssynergic defecation, however its mechanism of action is not known. The investigators hypothesize that biofeedback therapy enhances gut-brain-gut communication by altering cortical processing of information and improving cortically mediated neuromuscular function of the gut. The investigators' specific aims are; (1) To evaluate the afferent cortical evoked potentials in response to the electrical stimulation of the anorectum (i) before and after biofeedback therapy and (ii) compare responders with nonresponders. (2) To evaluate the corticofugal tracts (efferent) by recording the anal and rectal electromyographic responses following noninvasive lumbosacral and transcranial magnetic stimulation (i) before and after biofeedback therapy and (ii) compare responders with nonresponders.

The investigators hypothesize that biofeedback therapy enhances gut-brain-gut communication and alters cortical and neuromuscular function. The investigators' specific aims are to evaluate 60 patients with dyssynergia (i) before and after biofeedback therapy and (ii) compare responders with nonresponders by examining:

(A) The afferent cortical evoked potentials using electrical stimulation of the anus and rectum.

(B) The efferent cortical evoked potentials by lumbosacral and transcranial magnetic stimulation and recording the anal and rectal electromyographic responses.

ELIGIBILITY:
Inclusion Criteria:

* During the previous year, all patients must have experienced or reported at least two of the following symptoms for at least three months and with 25% of bowel movements (when not taking laxatives) (22):1) stool frequency of less than three/week, 2) passage of hard stools, 3) excessive straining, 4) a feeling of incomplete evacuation, 5)sensation of anorectal obstruction or blockage and 6) use of manual maneuvers to facilitate defecations (e.g., digital evacuation).
* No evidence of structural disease (excluded by colonoscopy/ b. enema and metabolic problem by lab tests.
* Patients on stable doses of antidepressants without anticholinergic effects will be included.
* Patient must be undergoing biofeedback treatment
* Patient must be right-handed

Exclusion Criteria:

* Patients taking drugs that are constipating, (e.g.; calcium channel antagonists will either be excluded or drug discontinued)
* Patients with comorbid illnesses; severe cardiac disease, chronic renal failure or previous gastrointestinal surgery except cholecystectomy and appendectomy.
* Neurologic diseases e.g.; head injury.epilepsy,multiple sclerosis, strokes, spinal cord injuries.
* Impaired cognizance (mini mental score of < 15) and/or legally blind.
* Pregnant or likely to conceive during the course of the study. Women with potential for pregnancy must be willing to use contraceptive measures during the study. Urinary pregnancy tests will be performed on such women prior to any radiologic procedures.
* Hirschsprung's disease.
* Alternating constipation and diarrhea (78).
* Ulcerative and Crohns colitis.
* Previous pelvic surgery, rectocele repair, bladder repair, radical hysterectomy.
* Rectal prolapse or anal fissure or anal surgery.
* Presence of metal in the skull, cranial cavity, back or hips.
* People who have a cardiac pacemaker, an implanted defibrillator, or a medication pump.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the afferent cortical evoked potentials using electrical stimulation of the anus and rectum (i) before and after biofeedback therapy and (ii) compare responders with nonresponders. | 2 visits of 3 hours each (3 months between 1st and 2nd visit)

CONTACTS AND LOCATIONS:
Overall Officials: Satish Rao, Md, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States